CLINICAL TRIAL: NCT00920231
Title: Computer Vision System for the Blind Veteran
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: C6731-R
Record Dates: First submitted 2009-06-11; First posted 2009-06-15 (Estimated); Results first posted 2015-04-02 (Estimated); Last update posted 2016-01-22 (Estimated); Status verified 2015-12

CONDITIONS: Blindness
MeSH Terms: conditions — Blindness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 initial system (Experimental): 8 blind subjects are asked to use a prototype computer vision system to determine the challenges facing computer vision based indoor navigation.
  Subjects are asked to travel through the hallways of a large hospital from the front entrance to a side entrance. The pathway consists of 9 segments including corners, four-way intersections, and doorways, and the total length of the route was approximately 200 meters. This challenging route was designed to stress the capabilities of the navigation system. It is a route that even sighted persons may find difficult to follow without practice. Pedestrian traffic was present throughout the route and lighting conditions could change in two of the segments where there were windows and doors.
  Interventions: Device: initial system
- Arm 2 modified system (Experimental): The system is redesigned in response to problems identified from the first phase of the study. The redesigned system is tested by a second set of 8 blind subjects in the same indoor path as used in Arm 1.
  Interventions: Device: modified system

INTERVENTIONS:
Device: initial system — The computer vision system is used to assist blind subject to navigate an extended path with multiple turns within a hospital setting.The initial prototype system would have been successfully tested for outdoor navigation and basic object recognition tasks.
  Arms: Arm 1 initial system
Device: modified system — The problems associated with the initial system were identified and modified. This modified system was tested with a second separate group of subjects. The redesigned system is used to assist blind subject to navigate the same extended path with multiple turns within a hospital setting.
  Arms: Arm 2 modified system

SUMMARY:
This is a feasibility study involving a small number of blind subject to evaluate the effectiveness of using a software and associated hardware components to assist the blind in identifying and locating objects of interests and to assist in way finding tasks. After the system has been successfully tested by the blindfolded engineers, it will be evaluated in a small number of blind subjects.

DETAILED DESCRIPTION:
This is primarily an engineering project to develop computer vision algorithms for an integrated system comprising of a laptop computer, webcam, gps, digital compass, microphone, and stereo earphones. The system will be voice controlled. The algorithm will be trained to identify and located objects and navigationally landmarks in real-time, previously selected by sighted developers. After the system has passed objective engineering milestones, blind subjects will be tested to determine whether the novel system will improve the ability of the blind to travel over a test course in a hospital setting.

ELIGIBILITY:
Inclusion Criteria:

* age 18 and over
* legally blind

Exclusion Criteria:

* decreased hearing
* unable to understand or follow instructions
* inability to walk and stand for 10 minutes

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2011-11; Primary Completion 2013-12 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cha-Min Tang, PhD MD, Principal Investigator — Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD
Locations (2):
- United States (2):
  - Atlanta VA Medical and Rehab Center, Decatur, Decatur, Georgia
  - Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD, Baltimore, Maryland

RESULTS

PARTICIPANT FLOW:
Groups:
- Initial Computer Vision System: a group of 8 blind subjects were tested with a prototype computer vision system build for outdoor navigation that relied on combination of GPS and location recognition for navigation information.
  the task was a wayfinding task starting from one point in the hospital and go to a point at another point in the hospital while navigating negotiating a number of turns over multiple corridors.
- Modified Computer Vision System: a second group of 8 blind subjects were tested with a modified computer vision system.
  same task as the initial group with improved computer vision algorithm.
Period: Overall Study
Arm/Group | Initial Computer Vision System | Modified Computer Vision System
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: a representative population for the VA of both sexes and ranging from 21 to 70. And they have a diverse set of reasons for blindness. But they all had sight once.
Groups:
- Initial System: a group of 8 blind subjects were tested with a prototype computer vision system build for outdoor navigation that relied on combination of GPS and location recognition for navigation information.
  the task was a wayfinding task starting from one point in the hospital and go to a point at another point in the hospital while navigating negotiating a number of turns over multiple corridors.
- Modified System: a second group of 8 blind subjects were tested with a modified computer vision system.
  same task as the initial group with improved computer vision algorithm.
- Total: Total of all reporting groups
Arm/Group | Initial System | Modified System | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 7 | 14
  >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Full Range); unit: years] — Initial system: 8 subjects with age range from 21 to 66; Modified system: 8 subjects with age range from 39 to 70
  years | 43 [21 to 66] | 52 [39 to 70] | 48 [21 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 5 | 3 | 8
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Device Failures Per Attempt to Complete a Navigation Course
Description: device failures were defined as any failure to provide correct location and direction information at thre appropriate time, resulting in a mistake that needed the initial prototype's ability to meet their travel needs at a good to excellent range.
Time Frame: The subject is given as much time as needed to complete the task
Measure: Mean (Standard Error); unit: number of device failures per attempt
Groups:
- Initial System: The subjects were asked to travel over a novel path in the hospital after given instructions how to reach the final destination. the computer vision system was used to provide additional information as when to turn and in what direction. the subjects were allowed to also use their white cane
- Modified System: a second group of 8 subjects were tested with a system that incorporated modifications identified by the first group using the initial prototype system.
Arm/Group | Initial System | Modified System
Number analyzed (Participants) | 8 | 8
number of device failures per attempt | 4.1 (1.2) | 2 (0.82)

2. Secondary Outcome: Ability to Meet the Subjective Travel Needs of the Blind Subject
Description: This is a subjective rating that incorporates user friendliness of the system and the specific needs of the subject. The subject is asked to rate whether the device meets his or her travel needs on a 1 to 7 scale with 1 being excellent and 7 being very poor.
Time Frame: no time limit
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Initial Prototype: The initial prototype is a system that has been successfully tested in outdoor navigation and successfully tested for simple object recognition.
- Modified System: this computer vision system incorporates the needed changes identified by the first group of subjects using the initial prototype system.
Arm/Group | Initial Prototype | Modified System
Number analyzed (Participants) | 8 | 8
units on a scale | 3.0 (0.30) | 2.3 (0.36)

ADVERSE EVENTS:
Groups:
- Arm 1: the blind subject is asked to locate a randomly placed object with the assistance of the webcam/laptop computer.
  computer vision: a webcam-laptop based system to assist the blind in locating objects and in way finding.
  No adverse events
- Arm 2: The subject without the assist device can only locate the object by groping and random searching with hands.
  No adverse events
Arm/Group | Arm 1 | Arm 2
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No